CLINICAL TRIAL: NCT05519956
Title: Elective Level Ib Irradiation in Nasopharyngeal Carcinoma Patients Based on the International Guidelines: an Open-label, Non-inferiority, Multicentre, Randomised Phase 3 Trial
Brief Title: Elective Level Ib Irradiation in Nasopharyngeal Carcinoma Patients Based on the International Guidelines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC008.1
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- level Ib-covering IMRT (Active Comparator): Patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II.
  Interventions: Radiation: level Ib-covering IMRT
- level Ib-sparing IMRT (Experimental): Patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II
  Interventions: Radiation: level Ib-sparing IMRT

INTERVENTIONS:
Radiation: level Ib-covering IMRT — Patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II.
  Arms: level Ib-covering IMRT
Radiation: level Ib-sparing IMRT — Patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II.
  Arms: level Ib-sparing IMRT

SUMMARY:
Currently, nasopharyngeal carcinoma (NPC) patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II will be recommended to receive level Ib-covering IMRT according to the International Guidelines. Our previous study, which retrospectively analyzed a cohort of 390 patients, indicated that it should be safe and feasible for patients who only had at least one of the above two radiological features. Thus, the investigators conduct this non-inferior phase 3, randomized trial to further determine the feasibility of sparing level Ib in patients who had level II involvement with ECE, and/or had a MAD of greater than 2cm in level II.

DETAILED DESCRIPTION:
Currently, nasopharyngeal carcinoma (NPC) patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II will be recommended to receive level Ib-covering IMRT according to the International Guidelines. Our previous study, which retrospectively analyzed a cohort of 390 patients, indicated that it should be safe and feasible for patients who only had at least one of the above two radiological features. Thus, the investigators conduct this non-inferior phase 3, randomized trial to further determine the feasibility of sparing level Ib in patients who had level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 2cm in level II.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed, non-metastatic nasopharyngeal carcinoma histologically confirmed by biopsy;
2. the following conditions: ① involvement of level II LNs with extracapsular extension(ECE); ② level II LNs involvement with maximum nodal axial diameter (MAD) greater than 2 cm;
3. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.

Exclusion Criteria:

1. level Ib involvement with positive pathological results;
2. submandibular glands (SMGs) involvement;
3. involvement of structures that drain to level Ib as the first echelon site (the oral cavity, anterior half of nasal cavity involvement);
4. previous malignancy or other concomitant malignant disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2022-09-16 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Regional relapse-free survival | 3 year
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.
level Ib recurrence rate | 3 year
  The level Ib recurrent rate will be calculated by the ratio of mumbers of patients relapsed in level Ib and the numbers of cases in the whole group.

SECONDARY OUTCOMES:
Local relapse-free survival | 3 year
  The local relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented local relapse or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Distant metastasis-free survival | 3 year
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented distant metastasis or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Overall survival | 3 year
  The overall survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Patient's quality-of-life: dry mouth | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: sticky saliva | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Lin, DR, Study Chair — Fujian Cancer Hospital